CLINICAL TRIAL: NCT00676949
Title: Phase I Study of Tumor Specific Potentiated Vaccine Therapy Using Cyclophosphamide Combined Epitope Peptide Cocktail for Progressive/Relapsed Solid Tumors(GI/Lung/Cervical Cancer)
Brief Title: Safety Study of Cancer Specific Epitope Peptides Cocktail for Cervical, GI, and Lung Tumors
Acronym: peptidevac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyushu University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Department of Advanced Molecular and Cell Therapy, Kyushu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KU-CY5peptides; 19-40 (Other: Kyushu University, Japan)
Record Dates: First submitted 2008-03-03; First posted 2008-05-13 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-04

CONDITIONS: Metastatic Tumors
Keywords: epitope peptide; cyclophosphamide; interleukin-2
MeSH Terms: conditions — Neoplasm Metastasis | interventions — LY6K protein, human; DEPDC1 protein, human; KIF20B protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): cyclophosphamide dose escalation, level 1:150mg/m2,level 2: 300mg/m2, level 3: 300mg/m2x2, with 5 kinds o tumor specific antigen peptides followed by low dose IL-2, 6 patients will be enrolled for each level.
  Interventions: Biological: 5 peptide vaccines of KOC1, TTK, CO16, DEPDC1, MPHOSPH1

INTERVENTIONS:
Biological: 5 peptide vaccines of KOC1, TTK, CO16, DEPDC1, MPHOSPH1 — 1mg each of 5 peptides with IFA. 4 weekly s.c. administration.
  Other Names: 5 peptide cocktail

SUMMARY:
The purpose of this study is to evaluate the clinical safety and efficacies of cyclophosphamide combined cancer specific epitope peptides cocktail for advanced/relapsed solid tumors including GI/lung/cervical cancers

DETAILED DESCRIPTION:
KOC1, TTK, CO16(URLC10), DEPDC1, MPHOSPH1 have been identified using genome-wide expression profile analysis by the use of cDNA microarray in the previous studies. The investigators have determined the HLA-A*2402 restricted epitope peptides respectively derived from KOC1, TTK, CO16(URLC10), DEPDC1, and MPHOSPH1 showed strong INF-gamma production when stimulated with the appropriate targets expressing the appropriate protein and HLA-A*2402. Furthermore, when vaccinated these peptides, specific CTLs were determined after the vaccination. Therefore the investigators focused on the prevention of further expansion of the solid tumors highly expressing these 5 proteins using these 5 peptides.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of unresectable or relapsed gastrointestinal, lung or cervical cancer patients
* performance status 0-1
* age between 20 and 80
* at least 4 weeks after previous therapy
* life expectancy more than 3 months
* permissible bone marrow, liver and renal function
* HLA-A2402
* no viral hepatitis, HIV or HTLV1

Exclusion Criteria:

* severe underlying disease
* pregnant or lactating women
* active brain metastasis
* uncontrollable infection
* under systemic corticosteroid or immune suppressant treatment
* history of allergy to epitope peptides or IFA

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
safety of the cyclophosphamide combined tumor specific epitope peptide cocktail | 2 years

SECONDARY OUTCOMES:
immunological efficacies and clinical efficacies of the cyclophosphamide combined tumor specific epitope peptides cocktail | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenzaburo Tani, MD,phD, Principal Investigator — Medical Institute of Bioregulation, Kyushu University
Locations (1):
- Kyushu University Hospital, Fukuoka, Fukuoka, Japan

REFERENCES:
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316